CLINICAL TRIAL: NCT06694584
Title: Study: Tea(m)Time - Strengthening the Team Resilience of Hospital Staff: A Quasi-experimental, Quantitative Pre-post Intervention Study
Brief Title: Study: Tea(m)Time - Strengthening the Team Resilience of Hospital Staff Through the Tea(m)Time Intervention
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Catholic University of Applied Sciences Mainz (Other)
Responsible Party: Principal Investigator, Ivonne Ledtermann, research assistant, Catholic University of Applied Sciences Mainz
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 23-034
Record Dates: First submitted 2024-10-24; First posted 2024-11-19 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Resilience, Psychological; Personnel, Hospital

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): Receives no intervention
- Tea(m)Time (Experimental): Tea(m)Time intervention: Tea(m)Time is divided into two phases, starting with the qualification of team leaders.
  The qualification is followed by the implementation of Tea(m)Time in the various teams.
  Interventions: Behavioral: Tea(m)Time

INTERVENTIONS:
Behavioral: Tea(m)Time — Tea(m)Time is divided into two phases, starting with the qualification of team leaders. This starts with knowledge transfer about healthy leadership, resilience, occupational health and safety, posture work, psychological empowerment, agile management and the role of the manager. The team leaders also learn various moderation/coaching techniques. The qualification is followed by the implementation of Tea(m)Time. The teams start each hour with self-reflection. This is followed by a stress assessment and prioritization. The teams then work on the problems identified and look for solutions together.
  Arms: Tea(m)Time

SUMMARY:
Employees in hospitals are exposed to various stressors and can be at risk of psychological stress. To counteract this, resilience programs are increasingly being offered. Most interventions focus on individual resilience. In this study, the focus is on the resilience of teams. For this reason, this research paper will focus on the Tea(m)Time intervention. Tea(m)Time is a health promotion intervention that combines the risk assessment of mental stress with a focus on team resilience. In order to generate knowledge about the Tea(m)Time intervention, this study aims to identify factors that promote and inhibit its implementation and mediate its effectiveness. The aim is to gain insights into the promotion of resilience in teams. The aim is to conduct the survey of the participants in the intervention group and the control group at three different points in time.

ELIGIBILITY:
Inclusion criteria:

* be at least 18 years old
* have sufficient knowledge of German
* are not on sick leave at time t0
* work in one of the planned clinics

Exclusion criteria:

* be younger than 18 years old
* do not have sufficient knowledge of German
* are on sick leave at time t0
* do not work in one of the planned clinics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-03-04 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
FITOR questionnaire (questionnaire on individual, team and organizational resilience) | t0 baseline, t1 6 months follow-up, t2 12 months follow-up
  Schulte, E.M. et al. (2021)

SECONDARY OUTCOMES:
Psychological empowerment | t0 baseline, t1 6 months follow-up, t2 12 months follow-up
  Schermuly, C.C. (2019)
Instrument to Measure the Culture for Psychological Empowerment in Organizations (IMPEC) | t0 baseline, t1 6 months follow-up, t2 12 months follow-up
  Schermuly, C.C. et al. (2022)
Organizational Commitment Questionnaire (OCQ-G) German version of the Organizational Commitment Questionaire | t0 baseline, t1 6 months follow-up, t2 12 months follow-up
  Maier, G.W. & Woschée, R. (2014) individual items were used
Assessment of Interprofessional Team Collaboration Scale II (AITCS-II) | t0 baseline, t1 6 months follow-up, t2 12 months follow-up
  Orchard C. (2015) individual items were used
Big-Five-Inventory-10 (BFI-10) | t0 baseline
  Rammstedt, B. et al. (2012)
The questionnaire to record the willingness to change (FEVER) | t0 baseline, t1 6 months follow-up, t2 12 months follow-up
  Hasler, G. et al. (2003). Testing of the German version of the University of Rhode Island Change Assessment Scale (URICA) individual items used and adapted
German standard version of the COPSOQ (Copenhagen Psychosocial Questionnaire) | t0 baseline, t1 6 months follow-up, t2 12 months follow-up
  FFAW (2023) individual items were used

CONTACTS AND LOCATIONS:
Overall Officials: Nadine Ungar, Dr., Principal Investigator — Professorship for Psychology in Healthcare
Locations (3):
- Germany (3):
  - Klinik Viktoriastift Bad Kreuznach, Bad Kreuznach
  - Geriatrische Fachklinik Rheinhessen-Nahe, Bad Kreuznach
  - Gesundheitszentrum Glantal, Meisenheim

IPD SHARING:
Plan to Share IPD: No